CLINICAL TRIAL: NCT02550418
Title: Open-label, Multi-centre, Proof of Concept Phase IIa Clinical Trial on the Efficacy and Tolerability of an 8 Week Oral Treatment With Once Daily 9 mg Budesonide in Patients With Active Ulcerative Colitis
Brief Title: Budesonide 9 mg Capsules in Active UC
Acronym: TOPICAL-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUX-3/UCA
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Budesonide (Experimental)
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide

SUMMARY:
The purpose of the trial is to evaluate the efficacy of an 8 week treatment with once-daily 9 mg budesonide in patients with active ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Men or women aged 18 to 75 years,
* Active ulcerative colitis, except proctitis limited to 15 cm ab ano, confirmed by endoscopy and histology,
* Established disease,

Exclusion Criteria:

* Crohn's disease, indeterminate colitis, ischaemic colitis, radiation colitis, microscopic colitis (i.e., collagenous colitis and lymphocytic colitis, incomplete microscopic colitis), diverticular disease associated colitis,
* Toxic megacolon or fulminant colitis,
* Colon resection,
* Evidence of infectious colitis (e.g., pathogenic bacteria or Clostridium difficile toxin in stool culture at screening),
* Malabsorption syndromes,
* Celiac disease,
* Bleeding hemorrhoids,
* Active peptic ulcer disease
* Other inflammatory or bleeding disorders of the colon and intestine, or diseases that may cause diarrhea or gastrointestinal bleeding,
* Hypertension, diabetes mellitus, osteoporosis, peptic ulcer disease, glaucoma, cataract, or infection if careful medical monitoring is not ensured,
* Any severe infectious disease (e.g., tuberculosis, AIDS),
* Severe co-morbidity substantially reducing life expectancy,
* History of colorectal cancer,
* History of cancer (other than colorectal) in the last 5 years, except for basal cell carcinoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission at final/withdrawal visit | 8 weeks treatment
  Clinical remission includes normalisation of stool frequency and absence of blood in stools

SECONDARY OUTCOMES:
Rate of endoscopic remission/improvement at final/withdrawal visit | 8 weeks treatment
Number of stools / bloody stools per week | 8 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Fellermann, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Fellermann K, Schiefke I, Racz I, Derova J, Jonaitis L, Wehrum S, Nacak T, Greinwald R. Efficacy and safety of prolonged release budesonide granules in mesalazine-refractory ulcerative colitis: A multi-centre Phase IIa study (TOPICAL-1). United European Gastroenterol J. 2020 Dec;8(10):1186-1195. doi: 10.1177/2050640620962632. Epub 2020 Oct 7. PMID 33028169